CLINICAL TRIAL: NCT02156297
Title: Sorafenib to Treat AML Patients With FLT3-ITD Mutation: a Non-interventional Cohort Study
Brief Title: Sorafenib to Treat FLT3-ITD AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: SZ3201
Record Dates: First submitted 2014-05-30; First posted 2014-06-05 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia; FLT3-ITD Mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Induction Group
- Consolidation Group
- Salvage Group
- Maintenance Group
- Alleviatitive Group

SUMMARY:
It is a prospective, non-interventional, open-label study, in order to observe the safety and response in FLT3-ITD mutation positive AML patients who receiving sorafenib as induction, consolidation, salvage, maintenance or alleviative treatment. The duration of the study from June 2014 through May 2019, with the recruitment duration from June 2014 to May 2017. The inclusion criteria is:

1. Definitely diagnosed as AML
2. FLT3-ITD mutation has been confirmed
3. Accepting the prescription of sorafenib

ELIGIBILITY:
Inclusion Criteria:

* Definitely diagnosed as AML
* FLT3-ITD mutation has been confirmed
* Accepting the prescription of sorafenib

Exclusion Criteria:

* Can not take drugs orally
* Can not follow the doctors' advices
* Other reasons that investigators considered as contra-indications for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed as AML with FLT3-ITD mutation and accepting the prescription of sorafenib.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2020-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | up to 2 years
Progress-Free Survival | up to 2 years

SECONDARY OUTCOMES:
Overall Survival | up to 2 years
Leukemia-Free Survival | up to 2 years
Median time to the onset of sorafenib resistance | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China